CLINICAL TRIAL: NCT00553618
Title: Adjuvant Interleukin2 (Proleukin)and 5-(3,3 Dimethyl-1-Triazeno) Imidazole-4-Carboxamide (DTIC) in Resected High-Risk Primary and Regionally Metastatic Melanoma
Brief Title: Adjuvant, Combined Interleukin 2 (Proleukin) and DTIC (Dacarbazine) in High-risk Melanoma Patients
Acronym: DTIC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Louisville (Other)
Collaborators: James Graham Brown Cancer Center (Other)
Responsible Party: Principal Investigator, Jason Chesney, Director, James Graham Brown Cancer Center, University of Louisville
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07.0008
Record Dates: First submitted 2007-11-01; First posted 2007-11-05 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Metastatic Melanoma
Keywords: Interleukin 2; Proleukin; DTIC; Dacarbazine; metastatic melanoma; adjuvant
MeSH Terms: conditions — Melanoma | interventions — aldesleukin; Dacarbazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Proleukin/DTIC Arm (Experimental): Adjucant proleukin and DTIC
  Interventions: Drug: Proleukin and Dacarbazine

INTERVENTIONS:
Drug: Proleukin and Dacarbazine — IL-2 (Proleukin), injected just under the skin, at a dose of 12 million units on days 1-4 for each of the six months of therapy.
  Dacarbazine, administered as an IV infusion through a freely flowing IV, at a dose of 750 mg, repeated every four weeks.
  Other Names: Proleukin, Dacarbazine

SUMMARY:
The purpose of this study is to see if the combination of the two cancer drugs, Dacarbazine (DTIC) and a low-dose of Proleukin (IL2), would provide a less toxic and more effective treatment for melanoma than currently available treatments for people with high-risk melanoma. Dacarbazine (DTIC) and Proleukin (IL2) are both FDA-approved drugs for the treatment of melanoma.

DETAILED DESCRIPTION:
The prognosis of patients with malignant melanomas that are greater than 4 mm deep or involve regional lymph nodes is poor, even after successful surgical removal. The concept of adjuvant therapy for melanoma is derived from the hypothesis that these therapies may kill micro-metastatic seeds of melanoma cells.

The rationale for this particular drug combination regimen is that melanoma cells may act as a vaccine from which to generate melanoma-specific T cell expansion by way of IL2 administration. In unpublished results, forty-two stage II and III melanoma patients were treated with this regimen at the University of Alabama with IRB approval. Analysis of relapse free survival and overall survival in patients treated with this combination suggested a small improvement in disease-free survival when compared to historical controls or another study whose patients had similar but not identical staging (median follow-up time of 30 months). Importantly, no unanticipated side effects were observed as a result of the combination of these two drugs (both of which are FDA-approved for use in melanoma patients).

ELIGIBILITY:
Inclusion Criteria:

* Patients must fulfill one of the following criteria:
* T4 NO MO - Deep primary melanoma (> 4.0 mm) with or without lymphadenectomy.
* T1-4 N1-3 MO - Primary melanoma with regional lymph node metastases found at lymphadenectomy or sentinel lymph node sampling, but clinically undetectable (occult).
* T1-4 N1-3 MO - Primary melanoma with clinically apparent (overt) regional lymph node metastases confirmed by lymphadenectomy.
* T1-4 N1-3 MO - Recurrence of melanoma at the proximal regional lymph node(s).
* Patients must have undergone a wide excision of the primary and, if >1mm in depth, have completed sentinel lymph node sampling or lymphadenectomy as is standard of practice. Patients must have confirmation of adequate surgical margins around the primary lesion (1 or 2 cm minimum, for primary lesions of 1-2 mm depth; 2 cm for primary lesions equal to or greater than 2 mm depth). When entering this study with recurrent regional lymph node disease, the patient must be enrolled no later than 90 days from the date of lymphadenectomy.
* For subungual melanomas a distal interphalangeal. amputation is required. For patients with regional lymph node recurrence, the same evidence for adequate margins around the primary are required as for patients at initial presentation.
* For safety reasons, patients must be of age between 18 and 85.
* Patients must have ECOG performance status 0-2.
* Patients must have WBC >3,000, platelet count >100,000, and hematocrit >33.
* Patients must have SGOT and bilirubin <2x normal; creatinine <2.3; BUN <33.
* Patients must have no active medical or psychiatric disorders requiring therapy that would prevent completion of the protocol.
* Patients must give written informed consent.

Exclusion Criteria:

* Patients for whom histopathologic examination of the primary or metastatic melanoma is not positive are ineligible.
* Patients who have clinical, radiological, laboratory, or pathological evidence of incompletely resected melanoma or any distant metastatic disease are ineligible.
* Patients with an active second cancer (except in situ cervical cancer, or basal or squamous skin cancer) are ineligible. Exceptions may be discussed with the principal investigator.
* Patients with organic brain syndrome or significant impairment of basal cognitive function or any psychiatric disorder that might preclude participation in the full protocol, are ineligible.
* Patients who have had prior adjuvant chemotherapy, immunotherapy, including preoperative infusion or perfusion therapy are ineligible.
* Patients with recurrent melanoma at regional lymph nodes must not have been previously entered into this study.
* Patients with more than one lymph node group involved are ineligible.
* Women of child bearing age who are not on adequate birth control are ineligible.
* Women who are pregnant or breast feeding are ineligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2007-08; Primary Completion 2025-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Relapse-free survival | The study duration is projected to be approximately 9 years

CONTACTS AND LOCATIONS:
Overall Officials: Jason A Chesney, MD, Principal Investigator — James Graham Brown Cancer Center, University of Louisville
Locations (1):
- James Graham Brown Cancer Center, Louisville, Kentucky, United States

REFERENCES:
- See also: James Graham Brown Cancer Center, Louisville, KY — http://www.browncancercenter.org